CLINICAL TRIAL: NCT01258855
Title: A Randomized Phase II Study of Sequential Biotherapy With Aflibercept and High Dose IL-2 Versus High Dose IL-2 Alone in Patients With Inoperable Stage III or Stage IV Melanoma: Efficacy and Biomarker Study
Brief Title: Aldesleukin With or Without Ziv-Aflibercept in Treating Patients With Stage III-IV Melanoma That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02498; NCI-2011-02498 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-107; CHNMC-PHII-107; CDR0000690654; 8628 (Other: City of Hope Comprehensive Cancer Center); 8628 (Other: CTEP); N01CM00038 (NIH); N01CM00070 (NIH); N01CM00071 (NIH); N01CM62209 (NIH); P30CA033572 (NIH); UM1CA186705 (NIH)
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Metastatic Melanoma; Recurrent Melanoma; Stage III Cutaneous Melanoma AJCC v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (ziv-aflibercept and aldesleukin) (Experimental): Patients receive ziv-aflibercept IV over at least 1 hour in weeks 1, 3, 5, and 7 (and in week 9 of course 1 only) and high-dose aldesleukin IV over 15 minutes every 8 hours for 5 days in weeks 1 and 3 (and in weeks 3 and 5 of course 1 only). Treatment repeats every 8 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance therapy comprising ziv-aflibercept IV on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Aldesleukin; Other: Laboratory Biomarker Analysis; Biological: Ziv-Aflibercept
- Arm II (aldesleukin) (Experimental): Patients receive high-dose aldesleukin IV over 15 minutes every 8 hours for 5 days in weeks 1 and 3. Treatment repeats every 4 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Aldesleukin; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Aldesleukin — Given IV
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Ziv-Aflibercept — Given IV
  Other Names: AFLIBERCEPT; AVE0005; Eylea; vascular endothelial growth factor trap; VEGF Trap; VEGF Trap R1R2; VEGF-Trap; Zaltrap
  Arms: Arm I (ziv-aflibercept and aldesleukin)

SUMMARY:
This randomized phase II trial studies how well aldesleukin with or without ziv-aflibercept works in treating patients with stage III-IV melanoma that cannot be removed by surgery. Aldesleukin may stimulate the white blood cells to kill cancer. Ziv-aflibercept may stop the growth of melanoma by blocking blood flow to the tumor. It is not yet known whether aldesleukin is more effective with or without ziv-aflibercept in treating melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the hypothesis that combination biotherapy with aflibercept (ziv-aflibercept) and high-dose (HD) interleukin (IL)-2 (aldesleukin) will improve the progression-free survival compared to HD IL-2 alone.

SECONDARY OBJECTIVES:

I. Evaluate the response rate (complete response [CR] + partial response [PR]) of aflibercept and HD IL-2 as assessed by Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1 and compare to results of HD IL-2 alone.

II. Evaluate the toxicities and tolerance of combination biotherapy with aflibercept and HD IL-2 and maintenance aflibercept alone in this patient population and compare to HD-IL2 alone.

III. Test the hypotheses related to the laboratory correlative studies. IV. Evaluate the overall survival of patients treated with aflibercept and HD IL-2 and HD IL-2 alone.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive ziv-aflibercept intravenously (IV) over at least 1 hour on day 1 of weeks 1, 3, 5, and 7 (and in week 9 of course 1 only) and high-dose aldesleukin IV over 15 minutes every 8 hours for 5 days in weeks 1 and 3 (and in weeks 3 and 5 of course 1 only). Treatment repeats every 8 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance therapy comprising ziv-aflibercept IV on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive high-dose aldesleukin IV over 15 minutes every 8 hours for 5 days in weeks 1 and 3. Treatment repeats every 4 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-4 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic melanoma (includes American Joint Committee on Cancer [AJCC] stage IV or advanced/inoperable stage III; also includes patients with a history of lower stage melanoma and subsequent recurrent metastatic disease that is either locally/regionally advanced/inoperable disease or distant metastases)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 10 mm with computed tomography (CT) scan or clinically (must be measurable with calipers) according to RECIST version 1.1
* Patients must be free of brain metastasis by contrast-enhanced CT/magnetic resonance imaging (MRI) scans within 4 weeks prior to enrollment; if known to have prior brain metastases, must not have evidence of active brain disease after definitive therapy (surgery, radiation therapy, or stereotactic radiosurgery) on two successive MRI evaluations at least 3 months apart (one of which is =< 4 weeks prior to starting the study drugs)
* A patient may be treatment naïve; however, up to two prior regimens for metastatic melanoma are allowed; prior adjuvant interferon (IFN)-alpha is allowed; no prior therapy with bevacizumab, aflibercept or interleukin-2 (IL-2)
* Patients must not have received systemic therapy or radiotherapy within the preceding 4 weeks; patients must have recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients must be at least 4 weeks from major surgery and have fully recovered from any effects of surgery, and be free of significant detectable infection
* For patients who have received prior anti-cytotoxic T-lymphocyte antigen (CTLA)4 monoclonal antibody therapy (ipilimumab or tremelimumab), there is a risk of bowel perforation with IL-2 therapy; therefore, for these patients if they have a history of colitis or diarrhea during anti-CTLA4 monoclonal antibody therapy, they should have a formal evaluation by a gastroenterologist and a colonoscopy should be considered to demonstrate the absence of active bowel inflammation before initiating IL-2 therapy on this protocol
* Life expectancy of greater than 3 months in the opinion of the investigator
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Karnofsky > 70%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within 1.5 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within 1.5 x institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine level above institutional normal
* Urine protein should be screened by urinalysis for urine protein creatinine ratio (UPCR); for UPCR > 1, a 24-hour urine protein should be obtained and the level should be < 500 mg
* Patients on full-dose anticoagulants (e.g., warfarin) with prothrombin time (PT) international normalized ratio (INR) > 1.5 are eligible provided that both of the following criteria are met:

  * The patient has an in-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin
  * The patient has no active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
* Forced expiratory volume (FEV) 1 > 2.0 liters or > 75% of predicted for height and age (pulmonary function test [PFTs] are required for patients over 50 years old or with significant pulmonary or smoking history)
* No evidence of congestive heart failure, symptoms of coronary artery disease, myocardial infarction less than 6 months prior to entry, serious cardiac arrhythmias, or unstable angina

  * Patients who are over 40 years old or have had previous myocardial infarction greater than 6 months prior to study entry or have significant cardiac family history (coronary artery disease [CAD] or serious arrhythmias) will be required to have a negative or low probability cardiac stress test (for example, thallium stress test, stress multi-gated acquisition scan [MUGA], stress echocardiography [echo], or exercise stress test) for cardiac ischemia within 8 weeks prior to registration
  * An echocardiogram should be performed at baseline in all patients; ejection fraction (EF) from baseline echocardiogram must be within the institutional limits of normal as determined by the reading cardiologist; if the baseline cardiac stress test incorporates an echocardiogram, then this will not need to be done again at baseline
* No history of cerebrovascular accident or transient ischemic attacks within the past 6 months
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 6 months after completion of study therapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Women should not be lactating and, if of childbearing age, should have a negative pregnancy test (beta-human chorionic gonadotropin [b-HCG] test; serum or urine, minimum sensitivity 25 IU/L or equivalent units of b-HCG) within two week of registration in the study
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with brain metastases should be excluded from this clinical trial except as noted above
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies, and patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to other agents used in the study
* Serious or non-healing wound, ulcer, or bone fracture
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment
* Patients with the following invasive procedures:

  * Major surgical procedures, open biopsy or significant traumatic injury within 28 days prior to day 1 therapy
  * Anticipation of need for major surgical procedures during the course of the study
  * Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to day 1 of therapy; central venous catheter placements are permitted to be completed 7 or more days prior to day 1 of therapy; however, peripherally inserted central catheter (peripherally inserted central catheter [PICC] or PIC line) may be placed at any time prior to or during therapy
* Patients with clinically significant cardiovascular or cerebrovascular disease:

  * History of cerebrovascular accident or transient ischemic attack within past 6 months
  * Uncontrolled hypertension, defined as blood pressure > 150/100 mm Hg or systolic blood pressure (BP) > 180 mm Hg if diastolic blood pressure < 90 mm Hg, on at least 2 repeated determinations on separate days within past 3 months
  * Myocardial infarction, coronary artery bypass graft (CABG) or unstable angina within the past 6 Months
  * New York Heart Association grade III or greater congestive heart failure, serious cardiac arrhythmia requiring medication, unstable angina pectoris within past 6 months
  * Clinically significant peripheral vascular disease within past 6 months
  * Pulmonary embolism, deep vein thrombosis (DVT), or other thromboembolic event within past 6 months
* History of tumor-related or other serious hemorrhage, bleeding diathesis, or underlying coagulopathy
* PT INR > 1.5 unless the patient is on full-dose warfarin
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients who have other current malignancies are not eligible; patients with other malignancies are eligible if they have been continuously disease free for > 5 years prior to the time of randomization; patients with prior history at any time of any in situ cancer, lobular carcinoma of the breast in situ, cervical cancer in situ, atypical melanocytic hyperplasia, or melanoma in situ are eligible; patients with a prior history of basal cell or squamous cell skin cancer are eligible; patients who have had multiple primary melanomas are eligible
* Patients must not have autoimmune disorders or conditions of immunosuppression that require current ongoing treatment with systemic corticosteroids (or other systemic immunosuppressants), including oral steroids (i.e., prednisone, dexamethasone) or continuous use of topical steroid creams or ointments or ophthalmologic steroids or steroid inhalers

  * If a patient had been taking steroids, at least 2 weeks must have passed since the last dose

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-01-18 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Tarhini, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (21):
- United States (21):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Virginia Cancer Center, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination Arm (Ziv-Afilbercept+HD IL2): Each course consisted of 2 cycles of HD IL2 at 600,000 IU/kg IV every 8 hours for up to 14 doses (1st cycle), followed by a period of 1 week rest and readmission for HD IL2 (2nd cycle). Ziv-aflibercept was given concurrently at 3 mg/kg IV every 2 weeks, starting 2 weeks prior to IL2 in course 1. In the absence of disease progression, maintenance ziv-aflibercept was given at 4 mg/kg every 2 weeks after completion of IL2
- Mono-therapy Arm (HD IL2 Alone): Patients received HD IL2 for a maximum of 3 courses (6 cycles)
Period: Overall Study
Arm/Group | Combination Arm (Ziv-Afilbercept+HD IL2) | Mono-therapy Arm (HD IL2 Alone)
Started | 55 | 29
Completed | 55 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Arm (Ziv-Afilbercept+HD IL2) | Mono-therapy Arm (HD IL2 Alone) | Total
Number analyzed (Participants) | 55 | 29 | 84
Age, Continuous [Median (Full Range); unit: years] | 55 [26 to 73] | 55 [31 to 74] | 55 [26 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 11 | 33
  Male | 33 | 18 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 54 | 28 | 82
  African American | 1 | 0 | 1
  Hispanic | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55 | 29 | 84

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: The time from the date of randomization until date of progression, death, or recurrence, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Arm (Ziv-Afilbercept+HD IL2) | Mono-therapy Arm (HD IL2 Alone)
Number analyzed (Participants) | 55 | 29
months | 6.9 [4.1 to 8.7] | 2.3 [1.6 to 3.5]
Statistical Analysis 1: Comparison: Combination Arm (Ziv-Afilbercept+HD IL2) vs Mono-therapy Arm (HD IL2 Alone); Test type: Other; p = 0.002, Log Rank

2. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: Until Death from any cause, up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Arm (Ziv-Afilbercept+HD IL2) | Mono-therapy Arm (HD IL2 Alone)
Number analyzed (Participants) | 55 | 29
months | 26.9 [14.4 to 63.6] | 24.2 [11.3 to 36.4]
Statistical Analysis 1: Comparison: Combination Arm (Ziv-Afilbercept+HD IL2) vs Mono-therapy Arm (HD IL2 Alone); Test type: Other; p = 0.43, Log Rank

3. Secondary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (RR) = CR + PR.
Time Frame: Up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Combination Arm (Ziv-Afilbercept+HD IL2) | Mono-therapy Arm (HD IL2 Alone)
Number analyzed (Participants) | 55 | 29
percentage of participants | 22 | 17

4. Secondary Outcome: Count of Participants With Adverse Events
Description: Count of the number of participants with grade 3 & 4 adverse events attributed to treatment agents. Events are graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Combination Arm (Ziv-Afilbercept+HD IL2) | Mono-therapy Arm (HD IL2 Alone)
Number analyzed (Participants) | 55 | 29
participants
  Anemia | 2 | 0
  Leukocytosis | 1 | 0
  Lymphocyte count decreased | 41 | 20
  Neutrophil count decreased | 2 | 0
  Platelet count decreased | 11 | 9
  Left ventricular systolic | 1 | 0
  Sinus tachycardia | 0 | 1
  Supraventricular tachycardia | 1 | 1
  Hypertension | 14 | 0
  Hypotension | 1 | 4
  Thromboembolic event | 2 | 1
  Fatigue | 5 | 3
  Fever and chills | 1 | 1
  Diarrhea | 0 | 1
  Oral mucositis | 0 | 1
  Nausea and vomiting | 2 | 2
  LFTs increased | 13 | 9
  Lipase increased | 0 | 2
  Confusion | 3 | 0
  Creatinine increased | 2 | 0
  Proteinuria | 6 | 0
  Urine output decreased | 8 | 7
  Dyspnea | 1 | 4
  Maculopapular rash | 1 | 0

5. Secondary Outcome: Progression-free Survival for Patients With High Vascular Endothelial Growth Factor (VEGF) Levels
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Median baseline measure for VEGF were used as the cut point for "low" vs "high" VEGF groups.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Arm (Ziv-Afilbercept+HD IL2) | Mono-therapy Arm (HD IL2 Alone)
Number analyzed (Participants) | 21 | 7
months | 8.7 [6.1 to 16.2] | 3.1 [1.5 to 7.4]
Statistical Analysis 1: Comparison: Combination Arm (Ziv-Afilbercept+HD IL2) vs Mono-therapy Arm (HD IL2 Alone); Test type: Other; p = 0.003, Log Rank

6. Secondary Outcome: Progression-free Survival for Patients With Low VEGF Levels
Description: as for outcome 5
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Arm (Ziv-Afilbercept+HD IL2) | Mono-therapy Arm (HD IL2 Alone)
Number analyzed (Participants) | 23 | 6
months | 6.9 [4.4 to 11.6] | 4.0 [1.2 to 6.9]
Statistical Analysis 1: Comparison: Combination Arm (Ziv-Afilbercept+HD IL2) vs Mono-therapy Arm (HD IL2 Alone); Test type: Other; p = 0.02, Log Rank

7. Other Pre Specified Outcome: 1-year Overall Survival Rate
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: Until Death from any cause, up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Arm (Ziv-Afilbercept+HD IL2) | Mono-therapy Arm (HD IL2 Alone)
Number analyzed (Participants) | 55 | 29
percentage of participants | 75.6 [64.5 to 88.6] | 66.8 [51.5 to 86.5]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded and graded throughout the study and until 30 days following the last dose of treatment agent.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Combination Arm (Ziv-Afilbercept+HD IL2) | Mono-therapy Arm (HD IL2 Alone)
All-Cause Mortality (participants affected / at risk) | 37/55 | 20/29
Serious Adverse Events (participants affected / at risk) | 28/55 | 7/29
Other Adverse Events (participants affected / at risk) | 55/55 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Arm (Ziv-Afilbercept+HD IL2) (N=55) | Mono-therapy Arm (HD IL2 Alone) (N=29)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Choledocholithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 15 (17) | 3 (3)
Lymphocyte count increased (Investigations) | 1 (12) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (4) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (9) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (2) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
splenic infarct (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Arm (Ziv-Afilbercept+HD IL2) (N=55) | Mono-therapy Arm (HD IL2 Alone) (N=29)
Anemia (Blood and lymphatic system disorders) | 40 (77) | 20 (39)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
hemoptysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
low carbon dioxide (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
red blood cells decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
white blood cells increased (Blood and lymphatic system disorders) | 7 (10) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (5)
Chest pain - cardiac (Cardiac disorders) | 2 (2) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Mobitz (type) II atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Mobitz type I (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 3 (4) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 39 (71) | 19 (61)
Supraventricular tachycardia (Cardiac disorders) | 1 (3) | 2 (3)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 3 (3) | 2 (2)
bigeminy ventricular arrhythemia (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 3 (3) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 1 (1)
Flashing lights (Eye disorders) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
diplopia (Eye disorders) | 2 (2) | 0 (0)
double vision (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 12 (15) | 7 (9)
Anal mucositis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 12 (16) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 40 (75) | 19 (31)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 6 (8) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric varices (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (3) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis nose (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 21 (27) | 6 (6)
Nausea (Gastrointestinal disorders) | 41 (85) | 20 (44)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 7 (8) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (3) | 0 (0)
Rectal mucositis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 30 (56) | 18 (40)
early satiety (Gastrointestinal disorders) | 1 (1) | 0 (0)
gum sensitivity (Gastrointestinal disorders) | 1 (1) | 0 (0)
mouth sores (Gastrointestinal disorders) | 1 (1) | 1 (1)
mouth ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
mouth ulcers (Gastrointestinal disorders) | 1 (1) | 0 (0)
mucosal edema (Gastrointestinal disorders) | 1 (1) | 0 (0)
oral mucosal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
tongue sensitivity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 40 (67) | 23 (44)
Edema face (General disorders) | 6 (9) | 6 (7)
Edema limbs (General disorders) | 25 (45) | 21 (30)
Edema trunk (General disorders) | 1 (1) | 2 (2)
Facial pain (General disorders) | 5 (5) | 0 (0)
Fatigue (General disorders) | 39 (75) | 22 (33)
Fever (General disorders) | 27 (46) | 19 (38)
Flu like symptoms (General disorders) | 4 (7) | 1 (1)
Infusion related reaction (General disorders) | 3 (3) | 0 (0)
Jaw Pain (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 8 (10) | 3 (4)
Non-cardiac chest pain (General disorders) | 2 (2) | 3 (3)
Pain (General disorders) | 5 (5) | 2 (4)
Rigors (General disorders) | 1 (1) | 1 (1)
Swollen Lips (General disorders) | 0 (0) | 1 (1)
edema LUE distal to PICC site (General disorders) | 1 (1) | 0 (0)
failure to thrive (General disorders) | 1 (1) | 0 (0)
night sweats (General disorders) | 1 (1) | 1 (1)
tongue edema (General disorders) | 0 (0) | 1 (1)
intra and extrahepatic biliary duct dila (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
seasonal allergies (Immune system disorders) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 3 (3) | 3 (4)
Oral Yeast (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Scrotal infection (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 4 (6) | 0 (0)
Skin infection (Infections and infestations) | 6 (6) | 1 (1)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Toe infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsilar abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 6 (8) | 0 (0)
Vaginal infection (Infections and infestations) | 2 (2) | 1 (1)
cellulitis (Infections and infestations) | 1 (1) | 0 (0)
only noted as bacteremia (Infections and infestations) | 0 (0) | 1 (1)
throat (Infections and infestations) | 1 (1) | 0 (0)
thrush (Infections and infestations) | 2 (2) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time pr (Investigations) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 31 (72) | 14 (19)
Alkaline phosphatase increased (Investigations) | 33 (84) | 16 (22)
Aspartate aminotransferase increased (Investigations) | 42 (93) | 16 (32)
Blood bilirubin increased (Investigations) | 37 (69) | 23 (42)
C Reactive Protein increased (Investigations) | 1 (1) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 2 (2) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 25 (48) | 8 (10)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Elevated Lactate dehydrogenase (Investigations) | 0 (0) | 1 (1)
Elevated lactate acid dehydrogenase (Investigations) | 1 (1) | 1 (1)
Elevated lactate dehydrogenase (Investigations) | 1 (1) | 0 (0)
Elevated neutrophil count (Investigations) | 1 (1) | 0 (0)
Elevated white blood cells (Investigations) | 1 (1) | 0 (0)
GGT increased (Investigations) | 2 (2) | 1 (1)
Hemoglobin increased (Investigations) | 2 (20) | 0 (0)
Hyperphosphatemia (Investigations) | 5 (8) | 0 (0)
INR increased (Investigations) | 4 (4) | 1 (1)
Increaesd LDH (Investigations) | 1 (1) | 0 (0)
LDH (Investigations) | 1 (1) | 0 (0)
LDH increased (Investigations) | 8 (12) | 4 (4)
LDH serum high (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 2 (3) | 2 (4)
Lymphocyte count decreased (Investigations) | 34 (69) | 18 (35)
Lymphocyte count increased (Investigations) | 13 (19) | 2 (2)
Neutrophil count decreased (Investigations) | 16 (39) | 12 (21)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Neutrphil count increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 46 (90) | 23 (46)
Platelet count increased (Investigations) | 4 (5) | 1 (1)
Serum amylase increased (Investigations) | 3 (7) | 0 (0)
Urine output decreased (Investigations) | 8 (10) | 7 (9)
Weight gain (Investigations) | 32 (48) | 18 (23)
Weight loss (Investigations) | 11 (40) | 3 (4)
White Blood Cells Increased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 23 (37) | 13 (21)
White blood cell increased (Investigations) | 3 (4) | 0 (0)
bicarbonate decreased (Investigations) | 2 (2) | 3 (3)
chloride increased (Investigations) | 0 (0) | 1 (1)
decreased appetite (Investigations) | 1 (1) | 0 (0)
decreased folic acid (Investigations) | 1 (1) | 0 (0)
decreased phosphorus (Investigations) | 2 (2) | 0 (0)
ele3vated phosphorus (Investigations) | 1 (1) | 0 (0)
elevated b natriuretic peptide (Investigations) | 1 (1) | 0 (0)
elevated lactate dehydrogenase (Investigations) | 9 (12) | 3 (3)
elevated platelet count (Investigations) | 1 (1) | 0 (0)
elevated white blood cells (Investigations) | 2 (2) | 1 (1)
generalized edema (Investigations) | 1 (1) | 0 (0)
increased LDH (Investigations) | 8 (8) | 0 (0)
increased PT (Investigations) | 1 (1) | 0 (0)
increased basophils (Investigations) | 0 (0) | 1 (1)
increased bilirubin, urine (Investigations) | 1 (1) | 0 (0)
increased chloride (Investigations) | 1 (1) | 0 (0)
increased eosinophils (Investigations) | 1 (1) | 1 (1)
increased phosphorous (Investigations) | 4 (5) | 0 (0)
increased phosphorus (Investigations) | 1 (1) | 0 (0)
increased platelets (Investigations) | 3 (3) | 0 (0)
increased thyroid stimulating hormone (Investigations) | 1 (1) | 0 (0)
increased white blood cells (Investigations) | 1 (1) | 0 (0)
lactate dehydrogenase (Investigations) | 2 (2) | 0 (0)
lactate dehydrogenase elevated (Investigations) | 4 (6) | 1 (1)
lactate dehydrogenase increased (Investigations) | 3 (4) | 1 (1)
lymhocyte count increased (Investigations) | 1 (1) | 0 (0)
neutrophil count increased (Investigations) | 3 (3) | 1 (1)
oliguria (Investigations) | 3 (5) | 2 (3)
platelet count increased (Investigations) | 5 (7) | 0 (0)
rigors (Investigations) | 1 (1) | 0 (0)
testosterone decreased (Investigations) | 1 (1) | 0 (0)
white blood cell increased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 19 (28) | 10 (11)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (10) | 6 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 22 (41) | 5 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 15 (22) | 5 (7)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (4) | 2 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 47 (106) | 24 (46)
Hypocalcemia (Metabolism and nutrition disorders) | 25 (42) | 13 (19)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (19) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 22 (38) | 10 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 41 (81) | 21 (38)
Hyponatremia (Metabolism and nutrition disorders) | 42 (83) | 19 (30)
Hypophosphatemia (Metabolism and nutrition disorders) | 37 (83) | 22 (42)
LDH Serum Increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
LDH Serum increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
LDH serum increased (Metabolism and nutrition disorders) | 11 (23) | 5 (6)
Obesity (Metabolism and nutrition disorders) | 1 (7) | 0 (0)
Phosphorus Increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
decreased bicarbonate (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
elevated chloride (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hyperphosphatemia (Metabolism and nutrition disorders) | 6 (11) | 0 (0)
low CO2 (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
low hemoglobin (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
phosphorus increasedf (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (16) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (18) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (19) | 2 (2)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pain at left clavicle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
rib pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
toe pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 11 (12) | 6 (7)
Dysgeusia (Nervous system disorders) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 23 (45) | 5 (5)
Lethargy (Nervous system disorders) | 3 (3) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Sinus pain (Nervous system disorders) | 4 (17) | 0 (0)
Somnolence (Nervous system disorders) | 2 (4) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 0 (0)
mental status changes (Nervous system disorders) | 1 (1) | 0 (0)
neurological episode NOS (Nervous system disorders) | 1 (1) | 0 (0)
paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
sleep disturbance (Nervous system disorders) | 1 (1) | 0 (0)
sleep disturbances (Nervous system disorders) | 1 (1) | 1 (2)
tingling, left foot (Nervous system disorders) | 0 (0) | 1 (1)
tingling, middle upper abdomen (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 7 (7) | 4 (5)
Anxiety (Psychiatric disorders) | 26 (38) | 14 (18)
Confusion (Psychiatric disorders) | 11 (12) | 8 (11)
Delirium (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 3 (3)
Hallucinations (Psychiatric disorders) | 5 (5) | 4 (5)
Insomnia (Psychiatric disorders) | 10 (10) | 7 (7)
Restlessness (Psychiatric disorders) | 1 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (3) | 3 (3)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 5 (5) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 25 (70) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 4 (9) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
decreased urine output (Renal and urinary disorders) | 1 (1) | 0 (0)
low urine output (Renal and urinary disorders) | 1 (1) | 0 (0)
renal insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)
urinary hesitancy (Renal and urinary disorders) | 2 (2) | 0 (0)
urinary pressure (Renal and urinary disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CO2 Decreased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 5 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 22 (26) | 14 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 (17) | 2 (2)
Odynophagia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 15 (20) | 6 (6)
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
dry nostrils (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
dry nostrils from O2 use (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 23 (26) | 15 (16)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema: chest and face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onychomalacia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 25 (30) | 17 (19)
Purpura (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (41) | 6 (7)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
callous, right hand (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
desquamation: hands, chest, foot, legs (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
desquamation: head and neck (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
erythema: thighs, legs, arms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
excoriation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
excoriation, groin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
peeling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
poison ivy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ruddy color, whole body (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
scrotal desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
white papules, lip (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
white spot on tonsil (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
xanthelasma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 5 (5) | 1 (1)
Flushing (Vascular disorders) | 10 (17) | 8 (12)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 29 (64) | 4 (6)
Hypotension (Vascular disorders) | 24 (40) | 22 (44)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT01258855/Prot_SAP_000.pdf